CLINICAL TRIAL: NCT00126230
Title: A Prospective Phase II Trial of Docetaxel-Samarium in Patients With Hormone-Refractory Advanced Prostate Cancer Who Achieve a Response or a Stabilization to Docetaxel-Estramustine
Brief Title: Trial of Docetaxel-Samarium in Patients With Hormone-Refractory Advanced Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAX-SAMAR
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: hormone-refractory advanced prostate cancer who achieve a response or a stabilization to docetaxel-estramustine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Samarium

INTERVENTIONS:
Drug: docetaxel and samarium

SUMMARY:
This is a prospective phase II trial of docetaxel-samarium in patients with hormone-refractory advanced prostate cancer who achieve a response or a stabilization to docetaxel-estramustine.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and less than 80 years
* Histologically-proven adenocarcinoma of the prostate
* Evidence of bone metastases and progressive, hormone-refractory, disease
* No previous chemotherapy
* No previous radiotherapy, except radiotherapy directed to the prostate and/or to a single bony lesion
* No previous carcinoma, except basal-cell carcinoma of the skin
* Adequate renal function: measured or calculated creatinine clearance > 60 ml/min
* Absolute granulocyte count ≥ 1,500/mm3, platelets ≥ 100,000 mm3, bilirubin ≤ 1.5 fold the upper normal value
* Signed informed consent.

Exclusion Criteria:

* Patients infected by the Human Immunodeficiency Virus (HIV)
* Patients who do not fit inclusion criteria

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2004-01

PRIMARY OUTCOMES:
Time to progression

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) response rate
Toxicity
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France